CLINICAL TRIAL: NCT02026908
Title: Prostatic Artery Embolization (PAE) for Treatment of Signs and Symptoms of Benign Prostatic Hyperplasia (BPH)
Brief Title: Prostatic Artery Embolization (PAE) for Treatment of Benign Prostatic Hyperplasia (BPH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Riad Salem, Professor of Radiology, Medicine and Surgery Chief, Section of Vascular and Interventional Radiology Director, Interventional Oncology Vice-Chairman, Image-Guided Therapy Department of Radiology Northwestern University, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 00081296; IDE G130133 (Other: FDA)
Record Dates: First submitted 2013-12-19; First posted 2014-01-03 (Estimated); Results first posted 2023-11-30 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2023-11

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
Keywords: Prostate Artery Embolization; PAE; Benign Prostatic Hyperplasia; BPH; Lower Urinary Tract Symptoms; LUTS
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prostate Artery Embolization (Experimental): There is only one arm of this study where patients receive Prostate Artery Embolization
  Interventions: Device: Prostate Artery Embolization

INTERVENTIONS:
Device: Prostate Artery Embolization — Procedure completed in Interventional Radiology includes a pelvic/prostate angiogram and embolization with Embosphere microspheres to slow/block blood flow to the prostate.

SUMMARY:
This is an open-labeled, non-randomized feasibility study to evaluate the safety of prostate artery embolization (PAE) for the treatment of lower urinary tract symptoms attributed to benign prostatic hyperplasia (BPH).

DETAILED DESCRIPTION:
This pilot study will be a single center, open labeled, non-randomized feasibility study to evaluate the initial safety of PAE for the treatment of symptomatic bladder outlet obstruction. 50 adult male subjects will be enrolled in this study. If eligible patients will undergo the prostate artery embolization procedure in the Interventional Radiology department. An angiogram of the prostate arteries will be done. Small beads called Embospheres will be injected into the prostate artery to slow blood flow to the prostate in the hope of providing relief with minimal side effects and complications, for lower urinary tract symptoms caused by BPH. After the procedure the patient will be followed at 4 weeks, 12 weeks, 6 months, 12 months post procedure and then annually for up to 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of LUTS secondary to BPH refractory to/contraindicated for medical treatment.
* Ability to understand and the willingness to sign a written informed consent
* Prostate volumes 40 - 200 gm. May include 30-39 gm if the subject has a long history of ineffective response to combination medical treatments (alpha-blocker and a 5-alpha reductase inhibitor) for at least 6 months
* Men ≥ 45 years of age
* IPSS symptom score > 13 and IPSS bother score > 2
* Peak flow rate Qmax≤ 12 with voided volume ≥125 cc

Exclusion Criteria:

* History of prostate or bladder cancer, pelvic radiation, untreated bladder stones,
* On alpha-blockers within the past 2 weeks unless on a stable dose of medication, with a stable urination pattern for 2 weeks prior to enrollment, and the willingness to stay on the same dose for the duration of the study, or until stopping criteria is met at the 12 month f/u visit, and or/part of a trial without catheter (TWOC) and patient is currently in Acute Urinary Retention (AUR)
* On 5-alpha reductase inhibitors within the past 6 months unless on a stable dose of medication with a stable urination pattern for 30 days prior to enrollment and the willingness to stay on the same dose for the duration of the study or until stopping criteria is met at the 12 month f/u visit .
* On phenylephrine, pseudoephedrine, imipramine, an anticholinergic or cholinergic medication within the past 2 weeks unless on a stable dose of medication with a stable urination pattern for 2 weeks prior to enrollment and the willingness to stay on the same dose for the duration of the study or until stopping criteria is met at the 12 month f/u visit .
* On estrogen, androgen, any drug producing androgen suppression, or anabolic steroids within the past 4 months unless on stable dose of medication for 30 days prior to enrollment and the willingness to stay on the same dose for the duration of the study.
* Daily use of a pad or device for incontinence required.
* Urethral strictures, renal insufficiency (i.e. creatinine > 1.8)
* Known primary neurologic conditions such as multiple sclerosis or Parkinson's disease or other neurological diseases known to affect bladder function.
* Neurogenic bladder, Hypotonic Bladder
* Prior treatment for urinary incontinence
* Penile prosthesis.
* Artificial urinary sphincter.
* Documented bacterial prostatitis within the past year.
* Active urinary tract infection (UTI) unless in case of regular catheter dependence and thought to represent colonization.
* History of chronic prostatitis within the last 1 year
* Known bleeding disorders (e.g. von willebrand disease (VWD))
* History of urethral strictures/bladder neck closure (BNC)
* Prior prostate procedures (e.g. Transurethral microwave therapy (TUMT), transurethral needle ablation of the prostate (TUNA), water-induced thermotherapy (WIT), transurethral resection of the prostate (TURP), photo-vaporization of the prostate (PVP))
* Prior treatment for overactive bladder (e.g. intravesical botox)
* Prostate Specific Antigen (PSA) > 4.0, < 10.0 unless documented negative prostate biopsy within past 2 years and is not thought to harbor prostatic malignancy in the clinical opinion of the primary or co-investigator.
* Enrolled in another treatment trial for any disease within the past 30 days
* Declines or unable to provide informed consent
* Condition precluding catheter-based intervention (ie occluded vessel, severe atheromatous disease)
* Any serious medical condition likely to impede successful completion of the study, such as certain mental disorders, uncontrolled diabetes, cardiac arrhythmias, cardiac disease including congestive heart failure, significant respiratory disease, or known immunosuppression.
* A history of rectal malignancy
* Prior surgical prostate intervention
* Interest in future fertility
* Allergy to Iodinated contrast agents not responsive to steroid premedication regimen
* Contraindication to Conscious sedation

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Riad Salem, MD MBA, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Salem R, Hairston J, Hohlastos E, Riaz A, Kallini J, Gabr A, Ali R, Jenkins K, Karp J, Desai K, Thornburg B, Casalino D, Miller F, Hofer M, Hamoui N, Mouli S. Prostate Artery Embolization for Lower Urinary Tract Symptoms Secondary to Benign Prostatic Hyperplasia: Results From a Prospective FDA-Approved Investigational Device Exemption Study. Urology. 2018 Oct;120:205-210. doi: 10.1016/j.urology.2018.07.012. Epub 2018 Jul 20. PMID 30036614

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were evaluated and followed by a multidisciplinary team including urology and interventional radiology.
Period: Overall Study
Arm/Group | Prostate Artery Embolization
Started | 45
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Prostate Artery Embolization
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 26
Age, Continuous [Mean (Full Range); unit: years] | 67 [47 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 42
  More than one race | 0
  Unknown or Not Reported | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 45
Length of BPH symptoms (years) [Mean (Full Range); unit: years] | 6.4 [1.5 to 21]
Mean Total Prostate Volume [Mean (Full Range); unit: cc] | 99 [30 to 214]
BUN (mg/dl) [Mean (Full Range); unit: mg/dl] | 19 [6 to 32]
Creatinine (mg/dl) [Mean (Full Range); unit: mg/dl] | 1.0 [0.4 to 17]
International Normalized Ratio (INR) [Mean (Full Range); unit: ratio] | 1.0 [0.9 to 1.1]
PSA (ng/ml) [Mean (Full Range); unit: ng/ml] | 3.4 [0.15 to 17.7]
percentage of Free PSA [Mean (Full Range); unit: percentage] — Measure Description: % Free PSA is the amount of the protein prostate-specific antigen (PSA) in the blood that is not attached to other proteins. It is compared with the amount of PSA in the blood that is attached to other proteins. The amount of free PSA is higher in men with benign prostatic hyperplasia (BPH).
  percentage | 24.1 [0.25 to 51.2]
Subjects with Abnormal Screening Urinalysis (RBCs) >4 per high Power field [Number; unit: participants] | 11
Subjects with Abnormal Screening Urinalysis (WBCs) >5 per high Power Field [Number; unit: participants] | 22

OUTCOME MEASURES:

1. Primary Outcome: The Primary Objective is to Evaluate the Safety of Prostate Artery Embolization (PAE) for the Treatment of Lower Urinary Tract Symptoms (LUTS) Attributed to Benign Prostatic Hyperplasia (BPH).
Description: The number and the severity of adverse events will be recorded to evaluate safety. Events will be reported by subjects and the severity of events will be graded using the following scale:
  Mild (grade 1): the event causes discomfort without disruption of normal daily activities Moderate (grade 2): the event causes discomfort that affects normal daily activities Severe (grade 3): the event makes the patient unable to perform normal daily activities or significantly affects his/her clinical status Life-threatening (grade 4): the patient was at risk of death at the time of the event Fatal (grade 5): the event caused death
Time Frame: 5 years
Measure: Number; unit: events
Arm/Group | Prostate Artery Embolization
Number analyzed (Participants) | 45
events
  Grade 1 AE Mild | 6
  Grade 2 AE Moderate | 10
  Grade 3 AE Severe | 1
  Grade 4 AE Life Threatening | 0
  Grade 5 AE Fatal | 0
Statistical Analysis 1: Comparison: Prostate Artery Embolization; Test type: Other — Paired T- test; p = 0.0001, t-test, 2 sided — P value was calculated with threshold of significance <0.05; p value = 0.05 — A p-value was calculated. Pretreatment (baseline) values for each parameter are compared to post-treatment values in a paired fashion

2. Secondary Outcome: Change in International Prostate Symptom Score (IPSS)
Description: Questionnaire-IPSS has 7 questions. Answer choices are as follows. The International Prostate Symptom Score (IPSS) can be utilized to measure the severity of lower urinary tract symptoms.
  It is a validated, reproducible scoring system to assess disease severity and response to therapy.
  The IPSS is made up of 7 questions related to voiding symptoms. Scores can range from 0-35 with 0 being the better outcome and 35 the worst outcome.
  Question 1-6 0-Not at all
  1. Less than 1 time in 5
  2. Less than half the time
  3. About half the time
  4. More than half the time
  5. Almost always
  Question 7 0-None 1-1 time 2-2 times 3-3 times 4-4 times 5-5 or more times
Time Frame: baseline, 4 weeks, 12 weeks, 6 months, 12 months, 2 years, 3 years, 4 years, 5 years
Population: Not all participants completed the questionnaire at all time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prostate Artery Embolization
Number analyzed (Participants) | 45
score on a scale
  Baseline: number analyzed (Participants) | 42
  Baseline | 23.6 (6.1)
  1 month follow up: number analyzed (Participants) | 42
  1 month follow up | 12 (5.9)
  3 month Follow up: number analyzed (Participants) | 41
  3 month Follow up | 10.2 (6.0)
  6 month follow up: number analyzed (Participants) | 41
  6 month follow up | 11.0 (7.6)
  12 month follow up: number analyzed (Participants) | 30
  12 month follow up | 12.4 (8.4)
  2 year follow up: number analyzed (Participants) | 21
  2 year follow up | 10.6 (6.78)
  3 year follow up: number analyzed (Participants) | 17
  3 year follow up | 8.3 (6.9)
  4 year follow up: number analyzed (Participants) | 16
  4 year follow up | 10.6 (6.5)
  5 year follow up: number analyzed (Participants) | 11
  5 year follow up | 11.1 (8.65)
Statistical Analysis 1: Comparison: Prostate Artery Embolization; Test type: Other — Paired t test; p = 0.0001, t-test, 2 sided — P value was calculated and a value of <0.05 was considered significant. A p-value was calculated. Comments: Pretreatment (baseline) values for each parameter are compared to post-treatment values in a paired fashion; p value = 0.05 — P value was calculated with threshold of significance <0.05

3. Secondary Outcome: Change in Quality of Life (QOL) Bother Question
Description: Questionnaire The total score ranges from 0-6 with 0 being the best outcome and 6 being the worst outcome.
  Questionnaire- answers choices are as follows:
  0- Delighted
  1. Pleased
  2. Mostly Satisfied
  3. Mixed about equality satisfied and dissatisfied
  4. Mostly Dissatisfied
  5. Unhappy
  6. Terrible
Time Frame: baseline, 4 weeks, 12 weeks, 6 months, 12 months, 2 years, 3 years, 4 years, 5 years
Population: Not all participants completed this score at all data points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prostate Artery Embolization
Number analyzed (Participants) | 45
score on a scale
  Baseline | 4.8 (0.9)
  1 month follow up | 2.6 (1.6)
  3 month follow up: number analyzed (Participants) | 44
  3 month follow up | 2.4 (1.6)
  6 month follow up: number analyzed (Participants) | 44
  6 month follow up | 2.3 (1.7)
  12 month follow up: number analyzed (Participants) | 31
  12 month follow up | 2.6 (1.6)
  2 year follow up: number analyzed (Participants) | 21
  2 year follow up | 1.9 (1.4)
  3 year follow up: number analyzed (Participants) | 17
  3 year follow up | 1.5 (1.2)
  4 year follow up: number analyzed (Participants) | 16
  4 year follow up | 2.2 (1.5)
  5 year follow up: number analyzed (Participants) | 11
  5 year follow up | 2.1 (1.4)
Statistical Analysis 1: Comparison: Prostate Artery Embolization; Test type: Other — Paired T test; p = 0.0001, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; p value = 0.05 — P value was calculated with threshold of significance <0.05

4. Secondary Outcome: Change in Benign Prostatic Hyperplasia (BPH) Impact Index
Description: Questionnaire The BPH Impact Index is to assess the impact of BPH symptoms on patient health and functioning. It is a self-administered questionnaire with 4 questions about urinary problems during the past month regarding physical discomfort, worry about health, how bothersome symptoms are, and whether the symptoms are interfering with doing usual activities.The BII is an evaluative index useful in measuring the magnitude of change in the impact of BPH-LUTS within a person over time.
  Scores range from 0-13 with 0 being the best outcome and 13 being the worst.
  Questionnaire- consists of 4 questions; answer choices are as follows Question 1: 0-none, 1-only a little, 2-some, 3-a lot Question 2: 0-none, 1-only a little, 2-some, 3-a lot Question 3: 0-not at all bothersome, 1- bothers me a little, 2-bothers me some, 3-bothers me a lot Question 4: 0-none of the time, 1- a little of the time, 2- some of the time, 3-most of the time, 4-all of the time
Time Frame: baseline, 4 weeks, 12 weeks, 6 months, 12 months, 2 years, 3 years, 4 years, 5 years
Population: Not all participants answered this questionnaire at all data points.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- There is Only One Arm for This Study.: All subjects underwent prostate artery embolization procedures.
Arm/Group | There is Only One Arm for This Study.
Number analyzed (Participants) | 45
score on a scale
  Baseline | 7.9 (2.4)
  1 month follow up | 3.8 (2.8)
  3 month follow up: number analyzed (Participants) | 43
  3 month follow up | 2.3 (2.5)
  6 month follow up: number analyzed (Participants) | 43
  6 month follow up | 2.5 (2.9)
  12 month follow up: number analyzed (Participants) | 31
  12 month follow up | 3.4 (3.1)
  2 year follow up: number analyzed (Participants) | 21
  2 year follow up | 2.1 (2.2)
  3 year follow up: number analyzed (Participants) | 17
  3 year follow up | 2.0 (2.2)
  4 year follow up: number analyzed (Participants) | 15
  4 year follow up | 2.2 (1.7)
  5 year follow up: number analyzed (Participants) | 11
  5 year follow up | 2.7 (2.1)
Statistical Analysis 1: Comparison: There is Only One Arm for This Study; Test type: Other — Paired T Test; p = 0.0001, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; p value = 0.05

5. Secondary Outcome: Change in Qmax (Peak and Total Void Volume at Each Follow-up Visit)
Description: Measure of urine flow rate. Q max = max flow rate. Peak Urine Flow (Qmax) from urodynamic assessments will be summarized comparing baseline to follow up measurements
Time Frame: baseline, 4 weeks, 12 weeks, 6 months, 12 months, 2 years, 3 years, 4 years, 5 years
Population: Low numbers of participants for the 12 month follow and later follow up visits are attributed to COVID when no visits were being made in person. Q max was not requied at the 6 month visit which is why no participates have data for this time point. no participants returned for the 5 year follow up for an in person visit.
Measure: Mean (Standard Deviation); unit: ml/second
Arm/Group | There is Only One Arm for This Study.
Number analyzed (Participants) | 45
ml/second
  Baseline: number analyzed (Participants) | 43
  Baseline | 5.8 (1.0)
  1 month follow up: number analyzed (Participants) | 43
  1 month follow up | 12.4 (6.8)
  3 month follow up: number analyzed (Participants) | 42
  3 month follow up | 15.3 (12.3)
  1 year follow up: number analyzed (Participants) | 25
  1 year follow up | 12.6 (12.1)
  2 year follow up: number analyzed (Participants) | 9
  2 year follow up | 12.4 (6.7)
  3 year follow up: number analyzed (Participants) | 3
  3 year follow up | 9.0 (6.7)
  4 year follow up: number analyzed (Participants) | 1
  4 year follow up | 3.1 (0)
Statistical Analysis 1: Comparison: There is Only One Arm for This Study; Test type: Other — Paired T test; p = 0.008, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; p value = 0.05 — P value was calculated and a value of <0.05 was considered significant. A p-value was calculated. Comments: Pretreatment (baseline) values for each parameter are compared to post-treatment values in a paired fashion

ADVERSE EVENTS:
Time Frame: Data was collected between the baseline visit up to 5 years post procedure date follow up. Baseline,4 weeks, 12 weeks, 6 months, 1 year, 2 year, 3 year, 4 year, 5 year.
Arm/Group | Prostate Artery Embolization
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

LIMITATIONS AND CAVEATS:
Since the pandemic started in 2020, annual visits were mostly preformed by completion of the IPSS questionnaire only, very few in person annual visits were completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT02026908/Prot_SAP_000.pdf